CLINICAL TRIAL: NCT01849601
Title: A Prospective, Multicenter and Single-arm Target Value Clinical Study on the Efficacy and Safety of Peripheral Balloon Dilatation Catheter in PTA Procedure
Brief Title: Effectiveness and Safety Study of Peripheral Balloon Dilatation Catheter in Percutaneous Transluminal Angioplasty(PTA) Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acotec Scientific Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: acotec-01
Record Dates: First submitted 2013-04-28; First posted 2013-05-08 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2012-11

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PTA catheter (Experimental)
  Interventions: Device: percutaneous transluminal angioplasty balloon catheter

INTERVENTIONS:
Device: percutaneous transluminal angioplasty balloon catheter
  Other Names: PTA catheter; trade name: Iris

SUMMARY:
The purpose of this study is to determine whether the peripheral balloon dilatation catheter (trade name: Iris) is safe an effective in PTA procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 yrs - 80 yrs.
* patients with iliac and / or femoral artery atherosclerotic lesions
* Rutherford grade of 1-5;
* Target lesion stenosis≥70% (visual estimation) (proportion of Trans-Atlantic Inter-Society Consensus(TASC) B, C and D grade lesions not less than 60% )
* Patients being able to understand the purpose of the test, and being volunteered to participate in and sign the informed consent.

Exclusion Criteria:

* Patients not suitable for receiving interventional surgeries of lower limb arteries for treatment;
* Patients require intervention of lesions besides unilateral iliac and femoral artery lesions at the same time;
* Patients have been involved in clinical trials of other drugs or medical devices within the past three months;
* Patient is unable or unwilling to participate in this trial;
* Patients with serious heart and brain, liver and other vital organs failure;
* Patients with life expectancy less than 6 months;
* Pregnant women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2012-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
technical success rate of PTA procedure | instant
  1. successfully pass lesion(s)
  2. successfully dilate lesion(s)( diameter of balloon reach at least 90% of the nominal diameter)
  3. successfully retrieve
  The definition of technical success rate of PTA procedure is that, all of the above 3 point are successful

SECONDARY OUTCOMES:
safety assessment | day 2 to day 10 after procedure or hospital discharge
  1. relevant balloon complications occurred during procedure(failure of balloon inflation, rupture of the balloon, failure of balloon deflation, failure of withdrawn, catheter fracture, etc.).
  2. Relevant major vascular complications occurred during procedure (rupture of blood vessels and acute vascular occlusion caused by dilation).

CONTACTS AND LOCATIONS:
Locations (1):
- Wei Guo, Beijing, China